CLINICAL TRIAL: NCT02415608
Title: A Phase 2 Study of Ibrutinib in Advanced Systemic Mastocytosis
Brief Title: Ibrutinib in Treating Patients With Advanced Systemic Mastocytosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Jason Robert Gotlib (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jason Robert Gotlib, Principal Investigator, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-31815; NCI-2014-02341 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEMMPD0021 (Other: OnCore); P30CA124435 (NIH)
Record Dates: First submitted 2015-03-24; First posted 2015-04-14 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Aggressive Systemic Mastocytosis; Mast Cell Leukemia; Systemic Mastocytosis
MeSH Terms: conditions — Mastocytosis, Systemic; Leukemia, Mast-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibrutinib 420 mg/day (Experimental): Participants receive ibrutinib daily on days 1 to 28, at 420 mg/day in 28-day cycles
  Interventions: Drug: Ibrutinib
- Ibrutinib 560 mg/day (Experimental): Participants receive ibrutinib daily on days 1 to 28, at 560 mg/day in 28-day cycles
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Given orally in 28-day cycles
  Other Names: Imbruvica; PCI-32765; BTK Inhibitor PCI-32765; CRA-032765

SUMMARY:
This phase 2 trial studies ibrutinib to see how well it works in treating patients with systemic (affecting the entire body) mastocytosis that has spread to other parts of the body and usually cannot be cured or controlled with treatment (advanced). Systemic mastocytosis is a disease in which too many mast cells (a type of immune system cell) are found throughout the body. Mast cells give off chemicals such as histamine that can cause flushing (a hot, red face), itching, abdominal cramps, muscle pain, nausea, vomiting, diarrhea, low blood pressure, and shock. Ibrutinib may stop the growth of mast cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

Evaluate the response rate to ibrutinib in patients with advanced systemic mastocytosis (SM) (aggressive systemic mastocytosis [ASM] or mast cell leukemia [MCL], or SM-associated hematologic non-mast cell disorder [AHNMD]) by the end of 6 cycles (6 months).

SECONDARY OBJECTIVES:

* Evaluate the tolerability and safety profile of ibrutinib in patients with advanced SM.
* Evaluate the pharmacokinetic (PK) profile of ibrutinib in a subset of patients with advanced SM.
* Evaluate changes in histopathology (blood and bone marrow) of patients with advanced SM in response to ibrutinib therapy.
* Evaluate changes in mastocytosis related symptom scores and quality-of-life (QOL) using a modified Myeloproliferative Neoplasm Symptom Assessment Form (MPNSAF).
* Evaluate the duration of response (DoR) and time to response (TTR).
* Evaluate progression-free survival (PFS) and overall survival.

OUTLINE:

Patients receive ibrutinib orally (PO) once daily (QD) on days 1 to 28. Treatment repeats every 28 days for up to 6 months in the absence of disease progression or unacceptable toxicity. Patients achieving an unconfirmed or confirmed clinical improvement (CI), partial response (PR), or complete response (CR) by the end of course 6 will be permitted to continue maintenance courses of ibrutinib on an ongoing basis until loss of response/progressive disease, or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 6 months thereafter.

ELIGIBILITY:
INCLUSION CRITERIA

* Diagnosis of systemic mastocytosis per 2008 World Health Organization (WHO) criteria. Those with advanced systemic mastocytosis (ASM); mast cell leukemia (MCL); or systemic mastocytosis-associated hematological clonal non-mast cell lineage disease (SM-AHNMD) required to have at least 1 organ damage finding
* Serum aspartate transaminase (AST) or alanine transaminase (ALT) ≤ 3.0 x upper limit of normal (ULN); if considered related to ASM/MCL ≤ 5 x ULN
* Estimated creatinine clearance ≥ 30 mL/min (Cockcroft-Gault)
* Total bilirubin ≤ 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin); if considered related to ASM/MCL ≤ 3 x ULN
* Female subjects must be of non-reproductive potential, or if of childbearing potential must have a negative serum pregnancy test upon study entry
* Must agree to use highly effective methods of birth control
* Written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 3
* Life expectancy > 12 weeks

EXCLUSION CRITERIA

* Received any investigational agent, chemotherapy, interferon-alpha, or 2-chlorodeoxyadenosine (2-CdA, cladribine) within 30 days prior to day 1; or monoclonal antibody ≤ 6 weeks prior to first administration of study treatment (patients with an AHNMD with progressive leukocytosis who require control of their counts are permitted to receive hydroxyurea)
* Diagnosis of AHNMD requiring immediate cytoreductive therapy or targeted drugs (eg, acute myeloid leukemia [AML])
* History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before the first dose of study drug, and at low risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* Concurrent systemic immunosuppressant therapy (eg, cyclosporine A, tacrolimus, etc., or chronic administration [> 14 days] of > 10 mg/day of prednisone) within 28 days of the first dose of study drug
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Systemic treatment for infection completed ≤ 14 days before the first dose of study drug
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4), grade 0 or 1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia
* Known bleeding disorders (eg, severe von Willebrand's disease) or severe hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Known history of human immunodeficiency virus (HIV) or
* Active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV)
* Major surgery within 4 weeks of first dose of study drug
* Any life-threatening illness, medical condition, or organ system dysfunction that could compromise the subject's safety or put the study outcomes at undue risk
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization
* Unable to swallow capsules or malabsorption syndrome
* Disease significantly affecting gastrointestinal function
* Resection of the stomach or small bowel
* Symptomatic inflammatory bowel disease
* Ulcerative colitis
* Partial or complete bowel obstruction
* Requires treatment with a strong cytochrome P450 (CYP) 3A4/5 inhibitor
* Lactating or pregnant
* Unwilling or unable to participate in all required study evaluations and procedures
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations)
* Known hypersensitivity to any excipient contained in the drug
* Received hematopoietic growth factor support within 14 days of day 1 of ibrutinib (Jehovah's witnesses may be given an erythropoiesis-stimulating agent before and during the trial in lieu of red blood cell transfusions but anemia and/or red blood cell (RBC) transfusion dependence cannot be used for response assessment in these patients)
* Presence of the factor interacting with poly(A) polymerase alpha (PAPOLA) and cleavage and polyadenylation specific factor 1 (CPSF1) (FIP1L1)-platelet-derived growth factor receptor, alpha polypeptide (PDGFRalpha) fusion even with resistance to imatinib (such patients are no longer defined as systemic mastocytosis by the WHO)
* Received any treatment with ibrutinib prior to study entry
* The concomitant use of warfarin or other vitamin K antagonists unless felt to be of significant clinical need; low molecular weight heparin or other anticoagulants may be used instead if anticoagulation is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-03; Primary Completion 2016-11-04 (Actual); Study Completion 2017-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gotlib, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibrutinib 420 mg/Day: Participants receive ibrutinib daily on days 1 to 28, at 420 mg/day in 28-day cycles
  Ibrutinib: Given orally
- Ibrutinib 560 mg/Day: Participants receive ibrutinib daily on days 1 to 28, at 560 mg/day in 28-day cycles
  Ibrutinib: Given orally
Period: Overall Study
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Full Range); unit: years] | 62.6 [61.6 to 78.5] | 76.8 [76.8 to 76.8] | 69.7 [61.6 to 78.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) is reported as the sum of the rates of participants achieving complete remission (CR), partial remission (PR), & clinical improvement (CI). A clinical response is a response with duration of ≥ 12 weeks.
  CR is defined as all 4 criteria:
  * No presence of compact neoplastic mast cell aggregates
  * Serum tryptase level < 20 ng/mL
  * Peripheral blood count remission defined as absolute neutrophil count (ANC) ≥1 x 10e9/L + normal differential, Hb ≥11 g/dL, & platelet count ≥100x10e9/L
  * Complete resolution of palpable hepatosplenomegaly & all biopsy-proven or suspected SM-related organ damage
  PR is defined as all 3 criteria with response duration ≥12 weeks, that is not CR or progressive disease:
  * ≥ 50% reduction in neoplastic mast cells
  * Serum tryptase level reduced ≥50%
  * Resolution of 1+ biopsy-proven or suspected systemic mastocytosis (SM)-related organ damage findings
  CI is defined as any improvement in any of the above measures.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day
Number analyzed (Participants) | 3 | 1
Participants | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, and reported as the number and percentage of participants having any adverse event; by each grade of adverse event; and by affected body systems.
Time Frame: 30 days
Population: All study participants are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day
Number analyzed (Participants) | 3 | 1
Participants
  Any Adverse event | 3 | 1
  Any Grade 1 Adverse Event (mild) | 3 | 1
  Any Grade 2 Adverse Event (moderate) | 3 | 1
  Any Grade 3 Adverse Event (severe) | 2 | 1
  Any Grade 4 Adverse Event (life-threatening) | 0 | 0
  Any Grade 5 Adverse Event (death) | 1 | 0
  Any Blood or Lymphatic System Disorder | 1 | 1
  Any Gastrointestinal Disorder | 1 | 1
  Any General Disorder | 3 | 1
  Any Infection or Infestation | 2 | 0
  Any Investigations | 1 | 0
  Any Metabolism or Nutrition Disorder | 1 | 1
  Any Musculoskeletal or Connective Tissue Disorder | 1 | 0
  Any Nervous System Disorder | 1 | 1
  Any Skin or Subcutaneous Tissue Disorder | 2 | 1
  Any Vascular Disorder | 1 | 0

3. Secondary Outcome: Ibrutinib Pharmacokinetics (PK)
Description: Plasma concentration-time profiles for each subject and mean plasma concentration-time profiles for each dose level will be plotted, plasma concentration data for ibrutinib at each time point will be summarized by descriptive statistics, and PK parameters such as maximum concentration (Cmax), minimum concentration, time at which the Cmax is reached, and area under the curve will be summarized with mean, geometric mean, medium, minimum, maximum, standard deviation, and coefficient of variation.
Time Frame: 28 days
Population: Because this study terminated with low total accrual, the funding sponsor elected not to analyze the samples for ibrutinib levels. There are no pharmacokinetics values on which to conduct the outcome analysis.
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change of Mast Cell Burden
Description: The change in the number of neoplastic mast cells in tissues (blood and/or bone marrow), ie, a measure of mast cell burden, will be assessed by immunophenotyping and/or immunohistochemistry (depending on patient and disease specifics) using mast cell markers, eg, CD25, CD30, CD117, tryptase, reticulin, Wright-Giemsa staining, and/or hematoxylin-eosin staining, in peripheral blood smears or bone marrow samples. For each participant, the data are used to collectively determine a single assessment for the number of mast cells present at baseline and after treatment. The outcome is reported as the median change in that level of mast cells, with full range, from baseline up to 2 years.
Time Frame: 2 years
Population: The result was only calculated for those participants for whom a post-treatment mast cell level could be determined.
Measure: Median (Full Range); unit: Percent reduction of mast cells
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day
Number analyzed (Participants) | 2 | 1
Percent reduction of mast cells | 47 [29 to 64] | 0 [0 to 0]

5. Secondary Outcome: Serum Tryptase Levels
Description: Serum tryptase level is a surrogate marker for the desired histopathologic response, ie, reduction in mast cell burden. Serum tryptase levels are reported as the median of the percent reduction, with full range, from baseline up to 2 years.
Time Frame: 2 years
Population: Results were determined for all participants.
Measure: Median (Full Range); unit: Percent reduction serum tryptase level
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day
Number analyzed (Participants) | 3 | 1
Percent reduction serum tryptase level | 30 [22 to 41] | 50 [50 to 50]

6. Secondary Outcome: Total Symptom Score (TSS)
Description: The totality of systemic mastocytosis was assessed by the total symptom score as measured by a Myeloproliferative Neoplasm Symptom Assessment Form modified for mast cell disorders [MPN-SAF (MCD)], and reported as the change in median score with standard deviation at baseline and 30 days. The MPN-SAF is a single, 27-question questionnaire that scores the following general measures on a scale of 0 (best) to 10 (worst): fatigue levels, effects of fatigue, satiety, pain, activity, concentration, dizziness, sleep, mood, anxiety, sexual function, itching, flushing, fever, weight loss, respiratory functions, diarrhea, lesions, and allergic reactions (some of these general terms may describe more than 1 assessment). The score on the MPN-SAF is the sum total of all 27 scores, and the range of scores is from a minimum of 0 (best; symptoms for all assessment absent) to a maximum of 270 (worst; score of 10 on all assessments).
Time Frame: 30 days
Population: Results were analyzed for all participants.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day
Number analyzed (Participants) | 3 | 1
score on a scale
  Cycle 1 Day ( baseline) | 56.0 (22.1) | 41 (NA) — Standard deviation can not be calculated on n=1.
  Cycle 2 Day 1 | 36.0 (15.0) | 41 (NA) — Standard deviation can not be calculated on n=1.

7. Secondary Outcome: Change in Quality of Life (QoL)
Description: The quality of life (QoL) component of the Myeloproliferative Neoplasm Symptom Assessment Form (MPNSAF) modified for mast cell symptoms, a scale of life quality ranking from 0 (best) to 10 (worst), was assessed at baseline and after 1 cycle of ibrutinib treatment (30 days), and reported as the median change in score with standard deviation.
Time Frame: 30 days
Population: Results were analyzed for all participants.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day
Number analyzed (Participants) | 3 | 1
score on a scale
  Cycle 1 Day (baseline) | 7.0 (1.0) | 6.0 (NA) — Standard deviation can not be calculated on n=1.
  Cycle 2 Day 1 | 7.0 (2.6) | 5.0 (NA) — Standard deviation can not be calculated on n=1.

8. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response (DoR) was assessed through 2 years of treatment, and reported as the median with standard deviation, with response duration censored at last response assessment in the event of death or progression not documented.
Time Frame: 2 years
Population: No participants achieved clinical response per protocol (minimum of any clinical improvement ≥ 12 weeks). On that basis, the overall duration of that response can not be determined.
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time-to-Response (TTR)
Description: Time-to-response (TTR) was assessed through 2 years of treatment, and reported as the median with standard deviation, censored at last response assessment in the event of death or progression not documented.
Time Frame: 2 years
Population: No participants achieved clinical response per protocol (minimum of any clinical improvement ≥ 12 weeks). On that basis, the time to achieve per-protocol clinical response can not be determined.
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Progression-free Survival (PFS)
Description: Participants were assessed for progression-free survival (PFS) from the start of treatment through 2 years of treatment. The outcome is reported as the number of participants who were alive without disease progression after 2 years of treatment.
Time Frame: 2 years
Population: Results were analyzed for all participants. Values were censored at the last assessment if the participant was lost-to-follow-up or otherwise did not have a 2-year assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day
Number analyzed (Participants) | 3 | 1
Participants | 0 | 0

11. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was assessed through 2 years of treatment, and recorded as the time from the start of treatment to either progression or death, with values censored at the last response assessment if the participant did not progress or die during that period. OS is reported as reported as the median with standard deviation.
Time Frame: 26 months
Population: The single patient receiving ibrutinib 560 mg/day was censored per protocol.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day
Number analyzed (Participants) | 3 | 0
months | 16.0 [6.4 to 25.6] |

ADVERSE EVENTS:
Time Frame: 26 months
Arm/Group | Ibrutinib 420 mg/Day | Ibrutinib 560 mg/Day
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib 420 mg/Day (N=3) | Ibrutinib 560 mg/Day (N=1)
Increased Aspartate aminotransferase (AST) (Investigations) | 1 (1) | 0 (0)
Increased alanine aminotransferase (ALT) (Investigations) | 1 (1) | 0 (0)
Increased total bilirubin (Investigations) | 1 (1) | 0 (0)
Increased alkaline phosphatase (Investigations) | 1 (1) | 0 (0)
Acute hepatitis A infection (Infections and infestations) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0)
Cryptococcal pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib 420 mg/Day (N=3) | Ibrutinib 560 mg/Day (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mouth sores (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue sensitivity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased fatigue (General disorders) | 3 (3) | 1 (1)
Cold symptoms (General disorders) | 1 (1) | 0 (0)
Edema, limbs (General disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron total, decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Basal cell carcinoma, scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythmateous rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin changes, fingertips (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Skin lesion, forearm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Increased flushing (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No